CLINICAL TRIAL: NCT03984344
Title: A Feasibility Trial of Theta Burst Stimulation in Anorexia Nervosa (AN)
Brief Title: Theta Burst Stimulation in Anorexia Nervosa
Acronym: ANTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KCLANTS19
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Anorexia Nervosa
Keywords: Theta Burst Stimulation; Neuromodulation; Psychiatric Disorders; Transcranial Magnetic Stimulation; Anorexia Nervosa; Eating Disorders
MeSH Terms: conditions — Anorexia Nervosa; Mental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of three treatment arms: continuous TBS or intermittent TBS or sham TBS.
Who Masked: Participant
Masking Description: Researcher unable to be blinded as stimulation site is dependent on the participants allocation to intermittent or continuous TBS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active iTBS (Experimental): iTBS will be delivered at 80% of resting motor threshold, consisting of a triplet of 50Hz bursts, repeated at 5Hz; 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 minutes and 9 seconds, to the left dorsolateral prefrontal cortex.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Active cTBS (Experimental): Continuous TBS will be delivered at 80% of RMT and will be applied as 600 pulses in a 40-second train of uninterrupted 50Hz bursts to the right dorsolateral prefrontal cortex.
  Interventions: Device: Continuous Theta Burst Stimulation
- Sham TBS (Sham Comparator): Sham stimulation will be given at the right or left dorsolateral prefrontal cortex (counterbalanced) for 40 seconds or 3 minutes and 9 seconds (counterbalanced), at the same frequency as active TBS (50Hz), however a sham coil will be used.
  Interventions: Device: Sham Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer active TBS.
  Other Names: iTBS
  Arms: Active iTBS
Device: Continuous Theta Burst Stimulation — The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer active TBS.
  Other Names: cTBS
  Arms: Active cTBS
Device: Sham Theta Burst Stimulation — The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer TBS using a sham Magstim coil.
  Other Names: Sham TBS
  Arms: Sham TBS

SUMMARY:
Anorexia Nervosa (AN) is a life-threatening eating disorder characterised by an intense fear of weight gain and disturbed body image, which motivates severe dietary restriction or other weight loss behaviours (e.g. purging). Treatment efficacy in adults with AN remains low: only a small percentage of individuals fully recover, and dropout rates are high. For adolescents with a relatively short term illness duration (under 3 years), family-based therapy has been associated with more favourable outcomes. However, for those adolescents with a longer illness duration (over 3 years), there are no specific treatments associated with positive long-term outcomes and these individuals are at risk of developing a severe and enduring form of the illness (SE-AN).

In part, treatment can be problematic due to ambivalence, which is reflected in poor take-up of certain treatments (e.g. pharmacological treatments that lead to weight gain) and high drop-out rates. Repetitive transcranial magnetic stimulation (rTMS) has demonstrated efficacy for treatment of AN in adults and improving treatment adherence. However, this has yet to be investigated in adolescents with AN.

This study will use a novel type of rTMS, theta burst stimulation (TBS), including intermittent TBS (iTBS) and continuous TBS (cTBS). TBS takes as little as a few minutes duration compared to the classical rTMS protocol which takes approximately 37.5 minutes. In addition, TBS has been found to produce longer after-effects of the induced plastic changes and has a lower stimulation intensity, which may therefore be more practical and potentially safer to administer in people with AN. Thus, the aim of this proof-of-concept trial is to obtain preliminary data on the safety and short-term (i.e. up to 24 hours) effects of a single session of iTBS and cTBS, compared to sham TBS, on reducing core symptoms of AN.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants over the age of 13
* BMI over 14 (for participants over the age of 18) or over 66% of the median BMI for age and gender (for participants under the age of 18)
* Right-handed
* Current Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of AN-restricting type (AN-R) or AN-binge/purge type (AN-BP) and an illness duration of 3 years or more
* Must have completed at least one adequate previous course of eating disorder treatment (e.g. one 6-month course of specialist outpatient therapy, specialist day-care or in-patient treatment for re-feeding)
* Participants under the age of 18 must have informed consent from parent(s)/carer(s)
* Must have approval from treating eating disorders clinician or general practitioner (GP) to participate

Exclusion Criteria:

* Having a history of head or eye injury
* Having a history of a neurological disease including previous seizures of any kind
* Having metallic implants anywhere in the head or body
* Being on a dose of any psychotropic medication that has not been stable for at least 14 days prior to participation in the study
* Taking antipsychotic medication
* Taking anti-convulsive medication
* Pregnancy or suspected pregnancy in female participants
* Having a current other major psychiatric disorder (e.g. major depressive disorder, substance dependence, schizophrenia or bipolar) needing treatment in its own right
* Excessive alcohol (>3 units per day, 5 days of the week) and/or cigarette consumption (>15 cigarettes per day)
* Severe abnormalities in the screening clinical blood sample
* An rTMS safety questionnaire and an MRI safety questionnaire will also be administered and if deemed not safe to deliver rTMS or undergo MRI scanning, people will be excluded on this basis.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes and differences between the 3 groups in core symptoms of AN from baseline to post-TBS | Baseline, within 1 hour after receiving [intermittent/continuous/sham] TBS, 24-hour follow-up
  Core symptoms of AN are computed by summing scores on three 10cm visual analogue scales (maximum score of 30) that assess levels of "urge to restrict", "feeling full", and "feeling fat". Participants are requested to indicate on this line a degree or level of experiencing the specific emotion or behavioural urge from "not at all" to "severe"

SECONDARY OUTCOMES:
Changes and differences between the 3 groups in heart rate from baseline to post-TBS | Baseline and within 1 hour after receiving [intermittent/continuous/sham] TBS
  Measures of heart rate (beats per minute) will be taken to assess cardiac safety of TBS in patients with AN
Changes and differences between the 3 groups in blood pressure from baseline to post-TBS | Baseline and within 1 hour after receiving [intermittent/continuous/sham] TBS
  Measures of blood pressure (millimetres of mercury; mmHg) will be taken to assess cardiac safety of TBS in patients with AN
Differences between the 3 groups in self-reported ratings of discomfort experienced during TBS | Within 1 hour of receiving [intermittent/continuous/sham] TBS
  Discomfort experienced during TBS will be measured using a 10cm visual analogue scales (maximum score of 10). Participants will be requested to indicate on this line a degree or level of discomfort experienced during TBS from "none" to "extreme discomfort"
Changes in performance on the Two-Step Sequential Learning Task from baseline to post-TBS | Baseline and within 1 hour of receiving [intermittent/continuous/sham] TBS
  Neuropsychological task measuring model-based and model-free reinforcement learning

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No